CLINICAL TRIAL: NCT03203941
Title: Autologous Cell Therapies for Cerebral Palsy-Chronic (ACT for CP) Individual Patient Expanded Access IND Protocol
Brief Title: ACT for CP Individual Patient Expanded Access IND Protocol
Status: No longer available | Type: Expanded Access
Sponsor: Charles Cox (Other)
Responsible Party: Sponsor-Investigator, Charles Cox, The George and Cynthia Mitchell Distinguished Chair in Neurosciences Director, Children's Program in Regenerative Medicine Professor, Department of Pediatric Surgery UTHealth McGovern Medical School at Houston, The University of Texas Health Science Center, Houston
Organization: The University of Texas Health Science Center, Houston (Other)
Other Study IDs: HSC-MS-17-0529
Record Dates: First submitted 2017-06-22; First posted 2017-06-29 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Cerebral Palsy
Keywords: Autologous Cord Blood Stem Cells
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Expanded Access Types: Individual, Treatment

INTERVENTIONS:
Biological: Autologous Cord Blood Stem Cells — This is an individual patient expanded access protocol.

SUMMARY:
Individual patient expanded access protocol for a child with cerebral palsy (CP) who has autologous umbilical cord blood available and who is ineligible to participate in other stem cell studies for children with CP.

DETAILED DESCRIPTION:
This protocol is part of an FDA Individual Patient Expanded Access IND submitted at the request of the parents of a child with cerebral palsy (CP) who is ineligible to participate in other stem cell studies. For this child, there are no other treatment options.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Charles S Cox, MD, Principal Investigator — UTHealth, McGovern Medical School at Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States